CLINICAL TRIAL: NCT07238933
Title: Neurological Events and Unforeseen Risks After Locoregional-anesthesia
Acronym: NEURAL
Status: Not yet recruiting | Type: Observational
Sponsor: Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva (Other)
Responsible Party: Sponsor
Other Study IDs: NEURAL
Record Dates: First submitted 2025-10-02; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Regional Anesthesia; Regional Anesthesia Block
Keywords: Nerve Injury; Pneumothorax; Local Anesthetic Systemic; Toxicity; Upper limb block; Lower limb block; Fascial plane block
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group of enrolled patients: Adult patients (≥18 years) undergoing single-shot upper limb, lower limb, or fascial plane regional anesthesia. All participants meeting inclusion criteria and providing informed consent will be enrolled consecutively.
  Interventions: Other: Observational assessment after regional anesthesia

INTERVENTIONS:
Other: Observational assessment after regional anesthesia — Adult patients undergoing single-shot regional anesthesia, including:
  Upper limb blocks - interscalene, superior trunk, supraclavicular, infraclavicular (coracoid, retroclavicular, costoclavicular), suprascapular (anterior, posterior), axillary, and superficial/intermediate/deep cervical plexus blocks.
  Lower limb blocks - lumbar, sacral, fascia iliaca (supra/infrainguinal), adductor canal, PENG, femoral, femoral triangle, sciatic (anterior, transgluteal, infragluteal, popliteal), nerve to vastus medialis, genicular, IPACK, common peroneal, ankle, and pudendal blocks.
  Fascial plane blocks - rectus sheath, ilioinguinal/iliohypogastric, TAP (standard/subcostal/midaxillary), ESP, serratus anterior (deep/superficial), parasternal intercostal (superficial/deep), interpectoral, transversalis fascia, rhomboid intercostal, retrolaminar, quadratus lumborum (anterior/lateral/posterior), paravertebral, intertransverse process, and pectoserratus blocks.

SUMMARY:
This is a multicenter, prospective, observational study aimed at determining the incidence of neurological and non-neurological complications following locoregional anesthesia procedures. The study will collect data on events such as nerve injury, hematoma, pneumothorax, and local anesthetic systemic toxicity.

DETAILED DESCRIPTION:
Locoregional anesthesia is generally considered safe, but rare neurological and systemic complications have been reported. Current data on the true incidence of these complications are limited and often derived from small sample sizes or registries. The NEURAL study aims to fill this knowledge gap by prospectively collecting data on complications following single-shot nerve blocks in the upper limb, lower limb, and fascial plane. In addition to incidence, the study will investigate potential risk factors for these complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Scheduled to undergo a single-shot nerve or fascial plane block.
* Ability to provide written informed consent.

Exclusion Criteria:

* Performance of more than one single-shot nerve or fascial plane block within the same anatomical region or sensory distribution during the same procedure.
* Use of continuous nerve or fascial plane catheter-based anesthesia.
* Presence of a language barrier that, in the investigator's judgment, would prevent adequate follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) undergoing single-shot locoregional anesthesia of the upper limb, lower limb, or fascial blocks.
Sampling Method: Non-Probability Sample
Enrollment: 3396 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Composite Complications Following Single-Shot Locoregional Anesthesia | From the time of the locoregional anesthesia procedure up to 30 days post-procedure (periprocedural and early postoperative period, with follow-up at 24 hours, 48 hours, 15 days, and 30 days).
  Incidence of any major complication - including nerve injury, hematoma requiring medical intervention, pneumothorax, or local anesthetic systemic toxicity (LAST) - following single-shot locoregional anesthesia. The rate is calculated as the number of procedures with at least one complication divided by the total number of procedures performed.

SECONDARY OUTCOMES:
Incidence of Complications in Upper Limb Nerve Blocks | From the procedure to 30 days post-procedure.
  Incidence of each complication type (nerve injury, hematoma, pneumothorax, LAST) following upper limb single-shot nerve blocks. Calculated as the number of events divided by the total number of upper limb procedures
Incidence of Complications in Fascial Plane Blocks | From the procedure to 30 days post-procedure.
  Incidence of each complication type (nerve injury, hematoma, pneumothorax, LAST) following fascial plane single-shot blocks.
(Predictor of Complications in Upper Limb, Lower Limb or Fascial Plane Blocks) Age | Baseline
  Measured in years
(Predictor of Complications in Upper Limb, Lower Limb or Fascial Plane Blocks) Gender | Baseline
  Using a dichotomic male/female framework
(Predictor of Complications in Upper Limb, Lower Limb or Fascial Plane Blocks) Body Mass Index | Baseline
  Calculated dividing a person's weight in kilograms by the square of their height in meters (BMI = weight ÷ height²) (kg/cm²)
(Predictor of Complications in Upper Limb, Lower Limb or Fascial Plane Blocks) Presence of comorbidities | Baseline
  Hypertension, diabetes, and central or peripheral neuropathies each expressed dichotomically as "Yes" (present) or "No" (absent).
(Predictor of Complications in Upper Limb, Lower Limb or Fascial Plane Blocks) Use of anticoagulant or antiplatelet therapy | Baseline
  Use of anticogulants and/or antiplatetets drugs expressed as a Yes or No
(Predictor of Complications in Upper Limb, Lower Limb or Fascial Plane Blocks) Use of sedative during the block procedure | Periprocedural
  Use of any sedative agents during the block procedure reported as a Yes or No
(Predictor of Complications in Upper Limb, Lower Limb or Fascial Plane Blocks) Pain at injection | Baseline
  Reported pain during the injection of local anesthetics expressed as a Yes or No
(Predictor of Complications in Upper Limb, Lower Limb or Fascial Plane Blocks) Ultrasound guidance | Periprocedural
  Use of ultrasound guidance to perform the block, measured with a "Yes" or "No" variable
(Predictor of Complications in Upper Limb, Lower Limb or Fascial Plane Blocks) Local anesthetic used to perform the block | Periprocedural
  Name, volume(ml) and dose(mg) of the local anesthetic used to perform the block
(Predictor of Complications in Upper Limb, Lower Limb or Fascial Plane Blocks) Adjuvants used to perform the block | Periprocedural
  Name, volume(ml) and dose(mcg) of the adjuvants used to perform the block

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro De Cassai Prof., MD, Principal Investigator — UOC Istituto di Anestesia e Rianimazione, Azienda Ospedale Università di Padova

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McLeod GA, Sadler A, Hales TG. Traumatic needle damage to nerves during regional anesthesia: presentation of a novel mechanotransduction hypothesis. Reg Anesth Pain Med. 2022 Jul 25:rapm-2022-103583. doi: 10.1136/rapm-2022-103583. Online ahead of print. PMID 35878962
- [Background] Gitman M, Fettiplace MR, Weinberg GL, Neal JM, Barrington MJ. Local Anesthetic Systemic Toxicity: A Narrative Literature Review and Clinical Update on Prevention, Diagnosis, and Management. Plast Reconstr Surg. 2019 Sep;144(3):783-795. doi: 10.1097/PRS.0000000000005989. PMID 31461049
- [Background] Neal JM, Barrington MJ, Brull R, Hadzic A, Hebl JR, Horlocker TT, Huntoon MA, Kopp SL, Rathmell JP, Watson JC. The Second ASRA Practice Advisory on Neurologic Complications Associated With Regional Anesthesia and Pain Medicine: Executive Summary 2015. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):401-30. doi: 10.1097/AAP.0000000000000286. PMID 26288034
- [Background] El-Boghdadly K, Wolmarans M, Stengel AD, Albrecht E, Chin KJ, Elsharkawy H, Kopp S, Mariano ER, Xu JL, Adhikary S, Altiparmak B, Barrington MJ, Bloc S, Blanco R, Boretsky K, Borglum J, Breebaart M, Burckett-St Laurent D, Capdevila X, Carvalho B, Chuan A, Coppens S, Costache I, Dam M, Egeler C, Fajardo M, Gadsden J, Gautier PE, Grant SA, Hadzic A, Hebbard P, Hernandez N, Hogg R, Holtz M, Johnson RL, Karmakar MK, Kessler P, Kwofie K, Lobo C, Ludwin D, MacFarlane A, McDonnell J, McLeod G, Merjavy P, Moran E, O'Donnell BD, Parras T, Pawa A, Perlas A, Rojas Gomez MF, Sala-Blanch X, Saporito A, Sinha SK, Soffin EM, Thottungal A, Tsui BCH, Tulgar S, Turbitt L, Uppal V, van Geffen GJ, Volk T, Elkassabany NM. Standardizing nomenclature in regional anesthesia: an ASRA-ESRA Delphi consensus study of abdominal wall, paraspinal, and chest wall blocks. Reg Anesth Pain Med. 2021 Jul;46(7):571-580. doi: 10.1136/rapm-2020-102451. PMID 34145070
- [Background] El-Boghdadly K, Albrecht E, Wolmarans M, Mariano ER, Kopp S, Perlas A, Thottungal A, Gadsden J, Tulgar S, Adhikary S, Aguirre J, Agur AMR, Altiparmak B, Barrington MJ, Bedforth N, Blanco R, Bloc S, Boretsky K, Bowness J, Breebaart M, Burckett-St Laurent D, Carvalho B, Chelly JE, Chin KJ, Chuan A, Coppens S, Costache I, Dam M, Desmet M, Dhir S, Egeler C, Elsharkawy H, Bendtsen TF, Fox B, Franco CD, Gautier PE, Grant SA, Grape S, Guheen C, Harbell MW, Hebbard P, Hernandez N, Hogg RMG, Holtz M, Ihnatsenka B, Ilfeld BM, Ip VHY, Johnson RL, Kalagara H, Kessler P, Kwofie MK, Le-Wendling L, Lirk P, Lobo C, Ludwin D, Macfarlane AJR, Makris A, McCartney C, McDonnell J, McLeod GA, Memtsoudis SG, Merjavy P, Moran EML, Nader A, Neal JM, Niazi AU, Njathi-Ori C, O'Donnell BD, Oldman M, Orebaugh SL, Parras T, Pawa A, Peng P, Porter S, Pulos BP, Sala-Blanch X, Saporito A, Sauter AR, Schwenk ES, Sebastian MP, Sidhu N, Sinha SK, Soffin EM, Stimpson J, Tang R, Tsui BCH, Turbitt L, Uppal V, van Geffen GJ, Vermeylen K, Vlassakov K, Volk T, Xu JL, Elkassabany NM. Standardizing nomenclature in regional anesthesia: an ASRA-ESRA Delphi consensus study of upper and lower limb nerve blocks. Reg Anesth Pain Med. 2024 Nov 4;49(11):782-792. doi: 10.1136/rapm-2023-104884. PMID 38050174
- [Background] Long B, Chavez S, Gottlieb M, Montrief T, Brady WJ. Local anesthetic systemic toxicity: A narrative review for emergency clinicians. Am J Emerg Med. 2022 Sep;59:42-48. doi: 10.1016/j.ajem.2022.06.017. Epub 2022 Jun 13. PMID 35777259